CLINICAL TRIAL: NCT00883285
Title: Incidence and Severity of Silent and Apparent Cerebral Embolism After Conventional and Minimal-invasive Transfemoral Aortic Valve Replacement
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Claas P. Naehle, Assistant Professor of Radiology, University Hospital, Bonn
Other Study IDs: 255/08
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Cerebral Stroke; Aortic Valve Disease
MeSH Terms: conditions — Stroke; Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: conventional aortic valve replacement
- 2: transfemoral aortic valve replacement
- 3: transapical aortic valve replacement

SUMMARY:
The purpose of this study is to compare the incidence of silent and apparent cerebral embolism between conventional and minimal-invasive transfemoral aortic valve repair.

DETAILED DESCRIPTION:
Patients undergoing aortic valve repair (AVR) are included prospectively into the study. AVR techniques include the conventional technique, the transfemoral and the transapical approach. Before the intervention CT of the chest is performed preoperatively to assess the degree of aortic and aortic valve calcification. Patients undergo MRI of the brain, including diffusion weighted imaging (DWI) and neurological assessment (NIHSS score) within 48 h before and after the procedure to assess occurrence of cerebral embolism.

ELIGIBILITY:
Inclusion Criteria:

* aortic valve replacement

Exclusion Criteria:

* contraindication to undergo MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic valve disease
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Silent cerebral embolism | 48 hours

SECONDARY OUTCOMES:
Apparent cerebral embolism | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bonn, Bonn, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Doerner J, Kupczyk PA, Wilsing M, Luetkens JA, Storm K, Fimmers R, Hickethier T, Eichhorn L, Naehle CP, Schild HH, Werner N, Nickenig G, Ghanem A. Cerebral white matter lesion burden is associated with the degree of aortic valve calcification and predicts peri-procedural cerebrovascular events in patients undergoing transcatheter aortic valve implantation (TAVI). Catheter Cardiovasc Interv. 2018 Mar 1;91(4):774-782. doi: 10.1002/ccd.27122. Epub 2017 May 26. PMID 28547872
- [Derived] Ghanem A, Kocurek J, Sinning JM, Wagner M, Becker BV, Vogel M, Schroder T, Wolfsgruber S, Vasa-Nicotera M, Hammerstingl C, Schwab JO, Thomas D, Werner N, Grube E, Nickenig G, Muller A. Cognitive trajectory after transcatheter aortic valve implantation. Circ Cardiovasc Interv. 2013 Dec;6(6):615-24. doi: 10.1161/CIRCINTERVENTIONS.112.000429. Epub 2013 Oct 15. PMID 24129642
- [Derived] Ghanem A, Muller A, Sinning JM, Kocurek J, Becker BV, Vogel M, Vasa-Nicotera M, Hammerstingl C, Schwab JO, Nahle CP, Thomas D, Wagner M, Grube E, Werner N, Nickenig G. Prognostic value of cerebral injury following transfemoral aortic valve implantation. EuroIntervention. 2013 Mar;8(11):1296-306. doi: 10.4244/EIJV8I11A198. PMID 23538093
- [Derived] Ghanem A, Muller A, Sinning JM, Kocurek J, Becker BV, Vogel M, Vasa-Nicotera M, Hammerstingl C, Schwab JO, Nahle CP, Thomas D, Wagner M, Grube E, Werner N, Nickenig G. Prognostic value of cerebral injury following transfemoral aortic valve implantation. EuroIntervention. 2012 Nov 22:20120710-05. Online ahead of print. PMID 23186915
- [Derived] Ghanem A, Muller A, Nahle CP, Kocurek J, Werner N, Hammerstingl C, Schild HH, Schwab JO, Mellert F, Fimmers R, Nickenig G, Thomas D. Risk and fate of cerebral embolism after transfemoral aortic valve implantation: a prospective pilot study with diffusion-weighted magnetic resonance imaging. J Am Coll Cardiol. 2010 Apr 6;55(14):1427-32. doi: 10.1016/j.jacc.2009.12.026. Epub 2010 Feb 24. PMID 20188503